CLINICAL TRIAL: NCT06088420
Title: Analgesic Efficacy of Erector Spinae Block , Quadratus Lumborum Block, and Intrathecal Morphine for Postoperative Pain Relief After Cesarean Section: A Randomized Study
Brief Title: Analgesic Efficacy of Different Nerve Blocks in Postoperative Cesarean Section
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Mamdouh Ekram, principal investigator., Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17101962
Record Dates: First submitted 2023-10-10; First posted 2023-10-18 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Population Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intrathcal Morphine Group (Active Comparator): Intrathecal morphine administration for post operative pain relief after cesarean section
  Interventions: Procedure: Intrathcal Morphine Group
- Quadratus Lumborum nerve block group (Active Comparator): Quadratus Lumborum nerve block administration for post operative pain relief after cesarean section
  Interventions: Procedure: Quadratus Lumborum nerve block(QL) group
- Erector Spinae nerve block group (Active Comparator): Erector Spinae nerve block administraion for post operative pain relief after cesarean section
  Interventions: Procedure: Erector Spinae nerve block (ESP)group

INTERVENTIONS:
Procedure: Intrathcal Morphine Group — intrathecal morphine (150 μg) in addition to standard spinal anesthetic drugs(10-12 mg 0.5% hyperbaric bupivacaine)
  Arms: Intrathcal Morphine Group
Procedure: Quadratus Lumborum nerve block(QL) group — intrathecal morphine (150 μg) in addition to standard spinal anesthetic drugs (10-12 mg 0.5% hyperbaric bupivacaine) + bilateral QL block by injecting 20 ml of 0.25% isobaric bupivacaine bolus with 4 mg ) dexamethasone as an adjuvant
  Arms: Quadratus Lumborum nerve block group
Procedure: Erector Spinae nerve block (ESP)group — intrathecal morphine (150 μg) in addition to standard spinal anesthetic drugs (10-12 mg 0.5% hyperbaric bupivacaine) + bilateral ESP block by injecting 20 ml of 0.25% isobaric bupivacaine bolus with 4 mg ) dexamethasone as an adjuvant
  Arms: Erector Spinae nerve block group

SUMMARY:
comparing analgesic efficacy of different nerve blocks on post operative cesarean sections.

DETAILED DESCRIPTION:
Analgesic efficacy of Erector Spinae, Quadratus Lumborum and Intrathecal Morphine for post operative pain relief after cesarean section,

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years old
* more or equal 37 weeks of gestation
* ASA 1,2
* Elective cesarean delivery

Exclusion Criteria:

* Patient refusal
* inability to cooperate with or understand the study
* local infection.
* bleeding disorder
* known anaphylaxis to any drug used in the trial
* ASA physical status more than 2
* emergency operations
* chronic opioid use (opioid use in the past 3 months)
* Neurologic deficit or disorder
* contraindication to regional anesthesia.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-10-15 (Actual); Primary Completion 2025-04-05 (Estimated); Study Completion 2025-04-05 (Estimated)

PRIMARY OUTCOMES:
Duration of analgesia until first analgesic request. | 24 hours .
  the time interval from immediate postoperative period until NRS reached 4

CONTACTS AND LOCATIONS:
Locations (1):
- Mahmoud Mamdouh Ekram, Asyut, Manfalout, Egypt

IPD SHARING:
Plan to Share IPD: No